CLINICAL TRIAL: NCT01486732
Title: FLT(3'-Deoxy-3'-[F-18]Fluorothymidine)-PET Activity Change After Allogeneic Umbilical Cord Blood Cell Therapy in Cerebral Palsy
Brief Title: FLT-PET Activity Change After Allogeneic Umbilical Cord Blood (UCB) Therapy in Cerebral Palsy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in obtaining specific isotope tracer
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, M.D., Associate Professor, Bundang CHA Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP FLT-PET
Record Dates: First submitted 2011-12-04; First posted 2011-12-06 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Umbilical Cord Blood; FLT-PET
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umbilical Cord Blood & Rehabilitation (Experimental): Allogeneic umbilical cord blood infusion and active rehabilitation
  Interventions: Biological: Umbilical Cord Blood Infusion; Other: Active Rehabilitation
- Placebo Umbilical Cord Blood & Rehabilitation (Active Comparator): Placebo Umbilical Cord Blood infusion and active rehabilitation
  Interventions: Other: Active Rehabilitation; Other: Placebo Umbilical Cord Blood

INTERVENTIONS:
Biological: Umbilical Cord Blood Infusion — The subjects will be undertaken allogeneic umbilical cord blood infusion intravenously or intraarterially under non-myeloablative immunosuppression.
  Other Names: Donated Umbilical Cord Blood Units from Affiliated Cord Blood Bank
  Arms: Umbilical Cord Blood & Rehabilitation
Other: Active Rehabilitation — All subjects should participate in active rehabilitation. They will receive two physical and occupational therapy sessions per day. Post discharge, each participant continued to receive rehabilitation therapy at least 3 days per week for additional 2.5 months.
Other: Placebo Umbilical Cord Blood — Placebo Umbilical Cord Blood that resembles cord blood in appearance was designed : 1.5 to 3 ml of the subject's own blood was collected and mixed with 15 to 20 ml of albumin
  Arms: Placebo Umbilical Cord Blood & Rehabilitation

SUMMARY:
This is randomized placebo-controlled trial to recognize new cell regeneration in the brain using FLT-PET.

DETAILED DESCRIPTION:
FLT(3'-Deoxy-3'-[F-18]Fluorothymidine) has been developed as a cell-proliferation tracer. In animal study, FLT-PET was used as a tool that enables imaging and measuring of proliferation in the brain, thus it detects activity of endogenous neural stem cells noninvasively. This study aims to assess cell proliferation activity changes in the brain after Umbilical Cord Blood (UCB)Therapy for Cerebral Palsy patients using FLT-PET.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy
* Abnormal muscle tone
* Gross Motor Function Classification System (GMFCS): I, II, III, IV, V
* Willing to comply with all study procedure

Exclusion Criteria:

* Medical instability including pneumonia or renal function at enrollment
* Presence of known genetic disease
* Presence of drug hypersensitivity which is related to this study remedy
* Poor cooperation of guardian,including inactive attitude for rehabilitation and visits for follow-up
* Decision by the principal investigator when there are unexpected events including brain surgery, that may affect the outcome

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of FLT-PET Activity Change | Baseline - 2 weeks
  Comparison of FLT-PET Activity Change between UCB group and Placebo group during 2 weeks: To compare differences in regional brain FLT-PET activity between groups and differences between pre- and post-therapy imaging data. The baseline and post-therapy data of each group will be compared using paired t-test statistics.

SECONDARY OUTCOMES:
Changes in Neurodevelopmental Outcome | Baseline - 2 weeks - 3 months
  Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Motor and Mental Scales (Higher score means better motor and mental function).
Changes in Standardized Gross Motor Function | Baseline - 2 weeks - 3 months
  GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 %, Higher score means better motor function).
Changes in Quality of Movement | Baseline - 2 weeks - 3 months
  GMPM (Gross Motor Performance Measure) as a standardized measurement tool for assessing quality of movement regarding 3 properties of 5 ones; alignment, coordination, dissociated movement, stability, and weight shift.

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea